CLINICAL TRIAL: NCT04168021
Title: Remote Ischemic Conditioning of the Human Brain in Dementia Patients (RICBDE): Protocol for a Crossover Non-pharmaceutical Intervention Study
Brief Title: Remote Ischemic Conditioning of the Human Brain in Dementia Patients
Acronym: RICBDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Greek Alzheimer's Association and Related Disorders (Other)
Responsible Party: Principal Investigator, Magda Tsolaki, Professor, Aristotle University Of Thessaloniki
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BrainIRC
Record Dates: First submitted 2019-11-10; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Mild Cognitive Impairment; Dementia; Intermittent Claudication
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Intermittent Claudication

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 90 individuals, baseline assessment before intervention (No Intervention): Baseline Cognitive status assessment
- Remote ischemic condition of the brain (Experimental): Intermittent claudication induction on a daily basis for 1 month
  Interventions: Behavioral: Leg ischemia
- Late cognitive assessment (No Intervention): Late cognitive status assessment 6 months later

INTERVENTIONS:
Behavioral: Leg ischemia — potential neuroprotection of ischemia/reperfusion of a peripheral organ or tissue against cerebral I/R injury
  Arms: Remote ischemic condition of the brain

SUMMARY:
The study investigates the incidence of remote ischemic conditioning in mild cognitive impairment and dementia patients

DETAILED DESCRIPTION:
The investigators will study the potential neuroprotection of ischemia/reperfusion (I/R) of a peripheral organ or tissue against cerebral I/R injury in people with mild cognitive impairment as well as early and middle stage dementia.

This crossover study will be held with individuals suffering from peripheral arteriopathy that can cause intermittent claudication after structured exercise, thus inducing extensive transient leg's ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild cognitive impairment
* Clinical diagnosis of mild dementia
* Clinical diagnosis of moderate dementia
* Peripheral arteriopathy

Exclusion Criteria:

* Clinical diagnosis of severe dementia
* Not being able to follow the exercise program for more than two days for any reason

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurements to Assess General Cognitive Function | Baseline, 1 and 6 months
  Change in Mini Mental State Examination (minimum value 10 - maximum value 30, higher scores mean a better outcome)
Neuropsychological Assessment | Baseline, 1 and 6 months
  Change Test (higher scores mean a better outcome)
Changes in Functional Cognitive State | Baseline, 1 and 6 months
  Global Deterioration Scale (values 1-7, higher scores mean a worse outcome)

SECONDARY OUTCOMES:
NeuroImaging | baseline, 1 month, 6 months
  Magnetic Resonance Imaging (MRI) (white matter hyperintensities volume)
Neurophysiology | Baseline, 1 month, 12 months
  Changes in Event-Related Potential (ERP) (oddball paradigm, auditory ERPs)
Electroencephalography recording | Baseline, 1 month, 6 months
  Changes in Electroencephalography (EEG), resting state

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available. Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices) will be shared. Study Protocol and Informed Consent Form will also be available. Data will be available (start and end dates) immediately following publication, No end date, with Investigations whose proposed use of the data has been approved by an independent review committee identified for this purpose, and for any purpose types of analysis.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available (start and end dates) immediately following publication, No end date
Access Criteria: To gain access, data requestors will need to sign a data access agreement.